CLINICAL TRIAL: NCT06038760
Title: Prospective Evaluation of AI R&D Tool in Adult Glioma and Other Primary Brain Tumours (PEAR-GLIO)
Acronym: PEAR-GLIO
Status: Terminated | Type: Observational
Why Stopped: Lack of funding
Sponsor: Ourotech, Inc. (Industry)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: PEAR-GLIO
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Brain Tumor; Glioma, Malignant; Ependymoma; Oligodendroglioma; Glioblastoma
Keywords: computer vision; cell culture; microtumor; functional testing; predictive biomarker; precision medicine; oncology; brain cancer
MeSH Terms: conditions — Brain Neoplasms; Glioma; Ependymoma; Oligodendroglioma; Glioblastoma; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor resections and blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trial Cohort: Patients with a solid primary brain tumor due to undergo surgery as standard of care
  Interventions: Procedure: Resection

INTERVENTIONS:
Procedure: Resection — Patients undergo a resection from a lesion, and give 40mL of blood

SUMMARY:
Pear Bio has developed a 3D microtumor assay and computer vision pipeline through which the response of an individual patient's tumor to different anti-cancer regimens can be tested simultaneously ex vivo. This study will recruit patients with primary brain tumors who are due to undergo surgery.

Oncologists will be blinded to treatment response on the Pear Bio tool (the assay will be run in parallel with the patient's treatment). The primary objective of this study is to establish the ex vivo model and confirm whether approved therapies exhibit their intended mechanism of action in the model. Secondary objectives include correlating test results to patient outcomes, where available.

DETAILED DESCRIPTION:
This is a multicenter, observational pilot study that aims to determine the feasibility of using the Pear Bio tool in patients with primary solid brain tumors.

Patients who are due to undergo clinically-mandated surgery will provide informed consent to donate excess tissue and a 40mL blood sample.

The samples will be tested on the Pear Bio tool while the patient receives their standard of care treatment. As such, for this study, the result from the Pear Bio tool will not be used to inform the choice of treatment and the treating oncologist will be blinded to the assay results.

The investigators will examine drug mechanism of action (MoA), differentiated response, and correlate that with outcomes seen in the patients treated in routine clinical practice.

ELIGIBILITY:
Inclusion:

1. Patient diagnosed with operable brain cancer, thought likely to be primary solid brain tumor on imaging (grade 2 - 3 meningioma; grade 1 - 4 tumors otherwise) or with histologically proven primary malignant solid brain tumor
2. Able to give written informed consent prior to admission to this study;
3. Female or male aged ≥18 years;
4. Patient consents to the use of their surgical sample and 40mL of whole blood for research purposes
5. Surgical sample and yields ≥0.4g for the study
6. Patient consents to providing histopathology data (e.g., confirmation of histological subtype as oligodendroglioma) and other pseudonymised health information including imaging, treatment and outcome data.

Exclusion:

1. Inoperable or biopsy only
2. Suspected lymphoma or myeloma, or grade 1 meningioma
3. Preoperative haemoglobin levels below 120g/L
4. Patients who have already received chemotherapy, targeted therapy, immunotherapy, or radiotherapy less than 30 days before date of surgery, unless as part of a clinical trial (requires per-patient sponsor approval)
5. Recurrence of cancer originating from a site other than the brain
6. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that may affect the interpretation of the results, render the patient at high risk from treatment complications or interferes with obtaining informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary solid brain tumor
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Differentiated ex vivo treatment response | 2 weeks
  Measurement of treatment response in the Pear Assay

SECONDARY OUTCOMES:
Progression-free survival correlation | 1 year
  The correlation between response in the Pear Bio system and PFS in patients

OTHER OUTCOMES:
Culture success rate of tumor cells | 1 week
  The percentage of cultures in which ≥70% of viable tumor cells encapsulated post-isolation on day 0 are still alive on day 3 in the control cultures (no treatment) compared to the number of tumor samples successfully accepted at the study central lab.
Culture rates success for immune cells | 1 week
  The percentage of cultures in which ≥70% of viable immune cells plated post-extraction on day 0 are still alive on day 3 in the control cultures (no treatment) compared to the number of blood samples successfully accepted at the study central lab.
Find correlations between ex vivo tumor culture or multi-omic biomarkers and real-world patient outcomes | 12 months
  To correlate Pear assay results, biomarkers and outcomes
Assess Pear Bio's assay ability to categorise patients for below average or above average overall survival (OS | 12 months
  Categorisation of patients into survival cohorts using the Pear assay
Assess the correlation of omics biomarkers to patient PFS, ORR and/or OS | 12 months
  Correlation between biomarkers and clinically relevant outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Matt Williams, FRCR PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pseudonymised data will be shared between study sites, such as treatment and outcome data for each patient. No publication will be made revealing individual patient data; only group-level data will be published.

REFERENCES:
- Available data/document: Study Protocol — https://www.pearbio.com/pearglio

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/60/NCT06038760/Prot_SAP_000.pdf